CLINICAL TRIAL: NCT02550054
Title: Erythropoietin in Premature Infants to Prevent Encephalopathy: A Multi-Centre Randomized Blinded Controlled Study of the Efficacy of Erythropoietin in China
Brief Title: Erythropoietin in Premature Infants to Prevent Encephalopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital, Fujian of China (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Guangzhou Women and Children's Medical Center (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Maternal and Child Health Hospital of Hubei Province (Other); The Maternal & Children Health Hospital of Dehong, Yunnan of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHFudanU_NNICU4; NCT02601872 (obsolete NCT alias)
Record Dates: First submitted 2015-09-04; First posted 2015-09-15 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth | interventions — Eosinophil Peroxidase; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental): Epo is administered 1000 U/kg, iv in 48 hours after premature birth, and at 48 hours interval for 3 doses per week. After 6 doses, Subcutaneously 3 doses per week until at corrected age of 34 weeks.
  Interventions: Drug: Epo
- Normal saline (Placebo Comparator): Normal saline is administered 5ml, iv at 3 to 6 hours after premature birth, and at 48 hours interval for 3 doses per week. After 6 doses, Subcutaneously 3 doses per week until at corrected age of 34 weeks.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Epo — Epo is administered 1000 U/kg, iv in 48 hours after premature birth, and at 48 hours interval for 3 doses per week. After 6 doses, subcutaneously 400 U/Kg per injection and 3 doses per week until at corrected age of 34 weeks.
  Other Names: Epoietin Beta
  Arms: Erythropoietin
Drug: Normal saline — Normal saline is administered 5ml, iv at 3 to 6 hours after premature birth, and at 48 hours interval for 3 doses per week. After 6 doses, Subcutaneously 3 doses per week until at corrected age of 34 weeks.
  Other Names: N/S solution
  Arms: Normal saline

SUMMARY:
The main goal of this trial is to investigate whether early administration of human erythropoietin (EPO) in preterm infants improves neurodevelopmental outcome at 18 months corrected age. This study is designed as randomized, double-masked, placebo controlled multicenter study involving at least 312 patients.

DETAILED DESCRIPTION:
EPO has been safely used for prevent preterm anemia and recent studies have shown the neuro-protective effect. Our hypothesis is that EPO could prevent preterm brain injury and reduce the rate of premature death and disability from encephalopathy. The aims of this study include: to investigate the safety and efficacy of EPO by using 1000u/kg higher than the dose of anemia treatment (250u/kg); to evaluate the effect of EPO on neurodevelopment in preterm infants; to detect biological and imaging indicators of EPO. Eligible premature infants will be enrolled in this double-blind, placebo-controlled randomized trial from the neonatal neurological intensive care unit (NNICU) at 7 Children's Hospital in 6 provinces of China. Subjects will be enrolled within the first 24 hours of life and randomly assigned to receive Epo or saline vehicle placebo. Standard NICU care will be provided to all subjects. Pharmacokinetic data, serial brain electrophysiologic and imaging exams, circulating inflammatory mediators, biomarkers and complications like polycythemia, neutropenia, thrombocytopenia, hypertension, sepsis, hemorrhage, seizure, necrotizing enterocolitis (NEC), persistent ductus arterious (PDA), apnea of prematurity, pulmonary haemorrhage, pulmonary hypertension, Prolonged blood coagulation time, retinopathy of prematurity (ROP), cardiac arrhythmia, major venous thrombosis, Renal failure treated with dialysis, pneumonia, pulmonary airleak and chronic lung disease will be collected at established time points during the study period. At 18 months corrected age, subjects will undergo a neurodevelopmental evaluation assessing for cerebral palsy, Bayley Scores of Mental Development Index (MDI) use.

ELIGIBILITY:
Inclusion Criteria:

1. Birthweight less or equal 1500 grams
2. Less than 32 weeks gestation at birth
3. Less than 48 hours of life at time of enrollment
4. Written informed consent of parent or guardian

Exclusion Criteria:

1. Intrauterine Growth Retardation
2. Severe Congenital Anomalies adversely affecting life expectancy or neurodevelopment
3. Genetic Metabolic Diseases
4. Seizures within first 24 hours of life
5. Severe neutropenia (ANC < 500 cells/microL) within first 24 hours of life
6. Polycythemia (Hct > 65%) within first 24 hours of life
7. Thrombocytopenia (platelets < 50K cells/microL) within first 24 hours of life
8. Hypertension (SBP > 100mmHg) without vasopressor support within first 24 hours of life
9. Microcephaly
10. Grade III-IV intracranial hemorrhage

Termination

1. Required by parent or guardian;
2. Polycythemia through blood transfusion can not be relieved
3. Oliguria（<0.5mL/kg/h for at least 24 hours）
4. Progression of azotemia
5. Pulmonary hypertension or Cardiac arrhythmia

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment(Bayley Scores) | At corrected age of 18 months
  To evaluate neurodevelopmental function via Bayley Scores of Infant Development Mental Development Index (BSID) and gain incidence of MDI<70(Severe) or MDI<85(Moderate).
Neurological Evaluation(GMFM-88 Scores) | At corrected age of 18 months
  To gain changes in standardized gross motor function using GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales, lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function).

SECONDARY OUTCOMES:
Brain Structural Alterations(MRI) | At corrected age of 9 months
  To compare changes in brain as measured by MRI in Epo treatment and control groups at 9 months.
Brain Structural Alterations(MRI) | At corrected age of 18 months
  To compare changes in brain as measured by MRI in Epo treatment and control groups at 18 months.
Intracranial Hemorrhage(MRI) | At corrected age of 9 months
  To compare changes in brain as measured by MRI in Epo treatment and control groups at 9 months.
Intracranial Hemorrhage(MRI) | At corrected age of 18 months
  To compare changes in brain as measured by MRI in Epo treatment and control groups at 18 months.
Brain Parenchyma Alterations(MRI) | At corrected age of 9 months
  To compare changes in brain as measured by MRI in Epo treatment and control groups at 9 months.
Brain Parenchyma Alterations(MRI) | At corrected age of 18 months
  To compare changes in brain as measured by MRI in Epo treatment and control groups at 18 months.
Somatosensory Evoked Potential | At corrected age of 9 months
  To compare changes in brain electrophysiology by SSEP at 36 weeks.
Somatosensory Evoked Potential | At corrected age of 18 months
  To compare changes in brain electrophysiology by SSEP at 18 months.
Visual Evoked Potential | At corrected age of 9 months
  To compare changes in brain electrophysiology by VEP at 36 weeks.
Visual Evoked Potential | At corrected age of 18 months
  To compare changes in brain electrophysiology by VEP at 18 months.
Brain Stem Auditory Evoked Potential | At corrected age of 9 months
  To compare changes in brain electrophysiology by BAER at 36 weeks.
Brain Stem Auditory Evoked Potential | At corrected age of 18 months
  To compare changes in brain electrophysiology by BAER at 18 months.
Incidence of complication | During treament period (in 34 weeks)
  To gain the incidence of Polycythemia, neutropenia, thrombocytopenia, hypertension, sepsis, intraventricular hemorrhage(IVH), periventricular leukomalacia(PVL), seizure, necrotizing enterocolitis (NEC), persistent ductus arterious (PDA), apnea of prematurity, pulmonary haemorrhage, pulmonary hypertension, Prolonged blood coagulation time, retinopathy of prematurity(ROP), cardiac arrhythmia, major venous thrombosis, Renal failure treated with dialysis, pneumonia, pulmonary airleak and chronic lung disease.
SDF-1 in Serum | At 34 weeks
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy of erythropoietin for hypoxic ischemic encephalopathy.
TNF-alpha in Serum | At 34 weeks
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy of erythropoietin for hypoxic ischemic encephalopathy.
IL-1 in Serum | At 34 weeks
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy of erythropoietin for hypoxic ischemic encephalopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Leuchter RH, Gui L, Poncet A, Hagmann C, Lodygensky GA, Martin E, Koller B, Darque A, Bucher HU, Huppi PS. Association between early administration of high-dose erythropoietin in preterm infants and brain MRI abnormality at term-equivalent age. JAMA. 2014 Aug 27;312(8):817-24. doi: 10.1001/jama.2014.9645. PMID 25157725
- [Background] Dame C, Langer J, Koller BM, Fauchere JC, Bucher HU. Urinary erythropoietin concentrations after early short-term infusion of high-dose recombinant epo for neuroprotection in preterm neonates. Neonatology. 2012;102(3):172-7. doi: 10.1159/000339283. Epub 2012 Jul 4. PMID 22776958
- [Background] Kuki I, Kawawaki H, Horino A, Inoue T, Nukui M, Okazaki S, Tomiwa K, Amo K, Togawa M, Shiomi M. [A clinical study on high-dose erythropoietin therapy for acute encephalopathy or encephalitis]. No To Hattatsu. 2015 Jan;47(1):32-6. Japanese. PMID 25803909
- [Background] Traudt CM, McPherson RJ, Bauer LA, Richards TL, Burbacher TM, McAdams RM, Juul SE. Concurrent erythropoietin and hypothermia treatment improve outcomes in a term nonhuman primate model of perinatal asphyxia. Dev Neurosci. 2013;35(6):491-503. doi: 10.1159/000355460. Epub 2013 Nov 1. PMID 24192275